CLINICAL TRIAL: NCT02658097
Title: A Phase II Trial of Pembrolizumab Sequentially Following Single Fraction Non-ablative Radiation to One of the Target Lesions, in Previously Treated Patients With Stage IV NSCLC
Brief Title: Pembrolizumab Alone or Sequentially Following Single Fraction Non-ablative Radiation to One of the Target Lesions, in Previously Treated Patients With Stage IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1516
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
Keywords: Lung Cancer; pembrolizumab; focal radiation; RT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Fraction Radiation Therapy (SFRT) + pembrolizumab (Experimental): 200mg Pembrolizumab by IV infusion on day 1 of each 3 week cycle. 8Gy will be given in a single fraction on the first day of treatment
  Interventions: Drug: Pembrolizumab; Radiation: Single Fraction Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg Pembrolizumab by IV infusion
Radiation: Single Fraction Radiation Therapy — 8Gy radiation therapy will be given in a single fraction on the first day of treatment
  Other Names: SFRT; RT

SUMMARY:
The goal of this clinical trial is to determine if low single palliative dose radiation to the lung cancer will improve your immune response against the tumor and if sequential treatment with pembrolizumab (the study drug) would offer superior results compared to pembrolizumab alone in participants with non-small cell lung cancer.

The purpose of this research is also to study whether there are any changes present in the DNA, RNA, and proteins of a participant's tumor or the blood cells that may contribute to a response to the study treatment or progression of cancer. This research may help researchers in the future to learn more about the causes, risks, treatments, or prevention of cancers or other health problems.

Participants will consent to a screening period, a core or treatment phase, and a post-study observation phase. During the screening phase, participants will undergo a series of tests to determine if they are eligible for the study. The core study period, or treatment period, will start with a single dose of radiation and then continue for the first eight treatments of pembrolizumab, approximately 24-28 weeks. Participants will have a new biopsy taken after two treatments of the study drug. Following the 24-28 week treatment cycle, if the cancer is responding to treatment, the participant's physician will continue to treat with pembrolizumab as a standard treatment. Following treatment, the post-study observation phase will monitor participant response to drugs and outcomes.

DETAILED DESCRIPTION:
The primary goal of this trial is to compare the efficacy of focal radiation (RT) to an index lesion as a way of enhancing the anti-tumor immune response to pembrolizumab to that of pembrolizumab alone. The primary efficacy endpoint is overall RECIST-defined response outside the radiation field.

Primary Objective: To determine the tumor responses outside the radiation field (abscopal effect) after radiation followed by pembrolizumab in metastatic NSCLC.

Secondary Objectives:

1. To determine the progression-free and overall survival in patients with NSCLC receiving pembrolizumab, who receive Single Fraction Radiation Therapy (SFRT)
2. To determine the safety and toxicity of the combination of SFRT and pembrolizumab
3. To examine potential predictive biomarkers in tumor samples and peripheral blood in patients treated with pembrolizumab and SFRT
4. To determine the local control of SFRT in the radiated lesion, when SFRT is given with pembrolizumab
5. To evaluate the induction of a T-cell response in patients with metastatic NSCLC treated with radiation and the effect of radiation

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor and primary investigator.
* Have a performance status of ≤1 ECOG Performance Scale.
* Demonstrate adequate organ function

  * Absolute neutrophil count (ANC) ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9g/dL
  * Serum creatinine or measured ≤1.5 times the upper limit of normal (ULN) or measured or calculated creatinine clearance ≥ 60 mL/min for subjects with creatinine levels >1.5 times the institutional ULN
  * Serum total bilirubin ≤ 1.5 X ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN or ≤ 5 times ULN for subjects with liver metastases
  * Albumin ≥ 2.5 mg/dL
* Have one measurable lesion of at least 1 cm outside the planned radiation field (defined as not receiving direct beam from any of the treatment portals).
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

* Male subjects of childbearing potential must agree to use an adequate method of contraception- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patient who have previously received radiation overlapping with the current planned radiation treatment fields are ineligible. Overlap is defined as any tissue falling within the direct path of both prior and current planned radiation fields.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patients with active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks and, have no evidence of new or enlarging brain metastases and also are off steroids 3 days prior to dosing with study medication. Stable brain metastases by this definition should be established prior to the first dose of pembrolizumab.
* Has had prior chemotherapy, within 2 weeks prior to study treatment. Patients on targeted therapy (tyrosine kinase inhibitor) may go on the study after 5 days off therapy.
* Patients who have not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to a previously administered agent.

  --Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C.
* Has received a live vaccine within 30 days of planned start of study therapy.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Pennell, MD, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
Age, Customized [Count of Participants; unit: Participants]
  40-49 years of age | 0
  50-59 years of age | 2
  60-69 years of age | 3
  70-79 years of age | 7
  80-89 years of age | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
Former Smoker [Count of Participants; unit: Participants] — Former smoker status of participants.
  Participants
    Former Smoker | 13
    Non-smoker | 0
Prior Treatment [Count of Participants; unit: Participants] — The number of prior treatments each participant were underwent before enrolling in this clinical trial.
  Participants
    1 prior treatment | 8
    2 prior treatments | 3
    3 prior treatments | 2
Types of prior treatments [Number; unit: number of prior treatments] — The types of prior treatments that participants received prior to enrolling in this clinical trial.
  number of prior treatments
    Carboplatin/Abraxane | 1
    Carboplatin/Pemetrexed | 5
    Cisplatin/Alimta | 1
    ETOPOSIDE / CARBOPLATIN 21 DAY | 1
    Maintenance Pemetrexed | 4
    Pemetrexed + Bevacizumab | 1
    Rucaparib | 2
    SBRT | 1
Sites of Metastatic Disease [Number; unit: number of sites] — The metastatic sites diagnosed in participant population.
  number of sites
    Bone site | 5
    Lung site | 1
    Lymph Nodes site | 8
Sites of Other Metastatic Disease [Number; unit: number of sites] — The other types of metastatic sites diagnosed in the patient population.
  number of sites
    Adrenal Gland site | 5
    Contralateral lung site | 7
    Kidney site | 1
    L supreaspinatus muscle site | 2
    Mediastinal LN site | 3
    Pleura site | 2
    Retoperitoneal LNs site | 2
    Rib site | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Each Response as Measured by RECIST 1.1
Description: The Best Overall Response is the best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The anti-tumor activity will be evaluated as an efficacy endpoints based on radiographic (CT or PET/CT). RECIST 1.1 will be applied for evaluation of tumor response. RECIST 1.1 criteria are as follows: Complete Response (CR) is defined as the disappearance of all lesions and pathologic lymph nodes; Partial Response (PR) is ≥ 30% decrease in sum of diameters with no new lesions, no progression of non-target lesions; Stable disease(SD) is defined as no PR - no progressive disease; and Progressive Disease (PD) is defined as ≥ 20% increase compared to smallest sum of diameters in study or progression of non-target lesions or new lesions.
Time Frame: From first visit to disease progression, up to 24 months after beginning treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
Participants
  Complete Response | 0
  Partial Response | 4
  Progressive Disease | 2
  Stable Disease | 5
  Not Evaluable | 2

2. Secondary Outcome: Median Time of Progression Free Survival
Description: Progression free survival, PFS is defined as the time from initiation of study drug post-SFRT, until the first documented, confirmed progression of disease. PFS will also be measured and report from the initiation of study drug, pre-SFRT.
Time Frame: From first visit to disease progression, up to 24 months after beginning treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
months | 3.5 [1.4 to NA] — N/A implies Not Reached; the upper side of the confidence interval has not been reached by the end of the follow up period.

3. Secondary Outcome: Median Time of Overall Survival
Description: Overall Survival, OS will be measure from the initiation of study therapy
Time Frame: From first visit to disease progression, up to 24 months after beginning treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
months | 9.2 [2.6 to NA] — N/A implies Not Reached; the upper side of the confidence interval has not been reached by the end of the follow up period.

4. Secondary Outcome: Number of Patients With Local Control of Disease With SFRT
Description: Local Control with SFRT: The target lesion selected for SFRT will be followed for local control. For the purpose of the study, local control will be defined as a complete response, partial response, or stable disease within the planning target volume.
Time Frame: From first visit to disease progression, up to 24 months after beginning treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
Participants | 9

5. Secondary Outcome: Duration of Local Control of Disease With SFRT
Description: Local Control with SFRT: The target lesion selected for SFRT will be followed for local control. For the purpose of the study, local control will be defined as a complete response, partial response, or stable disease within the planning target volume. The duration of local control will be measured from the time of SBRT treatment fraction.
Time Frame: From first visit to disease progression, up to 24 months after beginning treatment
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
months | 13 (11)

6. Other Pre Specified Outcome: Number of Patients With Pneumonitis
Description: For patients receiving SFRT to lung lesions, the development of grade 3 or greater pneumonitis that is probably or definitely attributable to either SFRT or pembrolizumab within the follow-up period will be monitored
Time Frame: From first visit to 30 days after disease progression, up to 25 months after beginning treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
Participants | 1

7. Other Pre Specified Outcome: Changes in PD-L1
Description: From first visit to disease progression, up to 25 months after beginning treatment. Median (95% CI) overall survival by PD-L1 status in months.
Time Frame: From first visit to 30 days post treatment, up to 25 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
Number analyzed (Participants) | 13
months
  Negative PD-L Status | 7.1 [4.7 to NA] — N/A implies Not Reached; the upper side of the confidence interval has not been reached by the end of the follow up period.
  Positive PD-L Status | 13 [2.1 to NA] — N/A implies Not Reached; the upper side of the confidence interval has not been reached by the end of the follow up period.

ADVERSE EVENTS:
Time Frame: Adverse events were collected up until 30 days after the final dose of study drug was administered to each participant.
Arm/Group | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 9/13
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Edema Cerebral (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Respitory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Fraction Radiation Therapy (SFRT) + Pembrolizumab (N=13)
Fatigue (General disorders) | 4 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Tracheal Mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
White blood cell decrease (Investigations) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 2 (3)
Creatinine increased (Investigations) | 2 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Dizziness (Nervous system disorders) | 2 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT02658097/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT02658097/ICF_001.pdf